CLINICAL TRIAL: NCT01415089
Title: Tailored Web-Based Intervention for Cancer Patients and Family Caregivers
Acronym: FOCUS-WEB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Wayne State University (Other); Barbara Ann Karmanos Cancer Institute (Other); Trinity Health Michigan (Other)
Responsible Party: Laurel Northouse PhD, Principal Investigator, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: R21CA138725 (NIH); R21CA138725 (NIH)
Record Dates: First submitted 2011-08-10; First posted 2011-08-11 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2013-10

CONDITIONS: Breast Cancer; Colorectal Cancer; Lung Cancer; Prostate Cancer
Keywords: Cancer; Quality of life; Family caregiver; Stress and coping; Web-based intervention; Communication
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Lung Neoplasms; Prostatic Neoplasms; Neoplasms; Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: FOCUS-Web — A 3-session individually tailored, interactive, web-based program providing support and education for cancer patients and one of their family caregivers.
  Other Names: FOCUS

SUMMARY:
The purpose of this pilot study is to develop a personalized, interactive, and web-based module for cancer patients and a family caregiver. The three-session module will be designed to help patients and family caregivers improve their communication and support.

DETAILED DESCRIPTION:
This R21 will be used to develop an individually tailored, interactive, web-based intervention for cancer patients (lung, colorectal, breast, prostate) and their family caregivers. This intervention is based on an efficacious, family-based program of care (the FOCUS Program) that has been tested previously in three large randomized clinical trials with positive outcomes for patients and their caregivers. In this R21 we will translate this primarily face-to-face, family-based program to an internet-based version.

The objectives are: Objective 1. To develop an individually-tailored, interactive, web-based and email-based, Family Involvement Module. We will conduct formative testing while developing the module using qualitative data obtained from four focus groups. We will conduct usability testing of the near final module with data obtained from qualitative interviews with patients and caregivers as they complete web-based task assignments using a "think aloud" protocol while they navigate the module. Objective 2. To conduct a Phase II study with cancer patients and their family caregiver (N = 40 dyads) using baseline (Time 1) and two-month follow-up assessments (Time 2). Between Times 1 and 2, all participants jointly will complete the web-based Family Involvement Module. We will determine the feasibility of delivering the web-based module and will obtain a process evaluation completed by study participants. Data will be obtained from three large cancer centers using established instruments, and analyzed with descriptive statistics and paired t-tests. Findings from this R21 will provide data that are essential to test this innovative, tailored, interactive web-based intervention with a larger sample in a R01.

ELIGIBILITY:
Inclusion Criteria:

* cancer patients with confirmed diagnosis of breast, colorectal, lung or prostate cancer
* early stage (I or II, diagnosed within past 2 to 12 months) OR advanced stage (III or IV, diagnosed or progressed within past 2 to 12 months)
* age 18 or older
* physically/mentally able to participate
* speak/read/write English
* have access to internet at home
* have a family caregiver willing to participate
* family caregivers must be age 18 or older, physically/mentally able to participate, able to speak/read/write English, identified by the patient as his or her primarily family caregiver, and have access to and willing to use the internet. "Family caregiver" is defined as the family member or significant other identified by the patient as his or her primary source of emotional or physical support during the current cancer experience and confirmed by the designated individual.

Exclusion Criteria:

* Family caregivers will be excluded from the study if they themselves have been diagnosed with cancer in the previous year or are receiving active treatment for cancer. This criteria was established so all dyads are managing effects of cancer in patients, not the family caregivers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2009-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Quality of life | Baseline (Time 1) and 2 months (Time 2)
  A preliminary assessment of the magnitude of the pilot intervention effects on patients' and family caregivers' level of quality of life (FACT-G Scale) will be conducted.

SECONDARY OUTCOMES:
Communication | Baseline (Time 1) and 2 months (Time 2)
  A preliminary assessment of the magnitude of the pilot intervention effects on patients' and family caregivers' level of communication (MIS Scale) will be conducted.
Dyadic support | Baseline (Time 1) and 2 months (Time 2)
  A preliminary assessment of the magnitude of the pilot intervention effects on patients' and family caregivers' level of dyadic support (Support Scale) will be conducted.
Self-efficacy | Baseline (Time 1) and 2 months (Time 2)
  A preliminary assessment of the magnitude of the pilot intervention effects on patients' and family caregivers' level of self-efficacy (CASE Scale) will be conducted.
Perceived benefits of illness | Baseline (Time 1) and 2 months (Time 2)
  A preliminary assessment of the magnitude of the pilot intervention effects on patients' and family caregivers' level of perceived benefits of illness (BOI Scale) will be conducted.
Emotional distress | Baseline (Time 1) and 2 months (Time 2)
  A preliminary assessment of the magnitude of the pilot intervention effects on patients' and family caregivers' level of emotional distress (POMS Scale) will be conducted.
Satisfaction with intervention | 2 months after baseline survey (Time 2)
  An assessment of the patients' and family caregivers' level of satisfaction with the intervention (Process Evaluation) will be conducted.

CONTACTS AND LOCATIONS:
Overall Officials: Laurel Northouse, PhD, Principal Investigator — University of Michigan School of Nursing
Locations (3):
- United States (3):
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan

REFERENCES:
- [Background] Zulman DM, Schafenacker A, Barr KL, Moore IT, Fisher J, McCurdy K, Derry HA, Saunders EW, An LC, Northouse L. Adapting an in-person patient-caregiver communication intervention to a tailored web-based format. Psychooncology. 2012 Mar;21(3):336-41. doi: 10.1002/pon.1900. Epub 2011 Jan 23. PMID 21830255
- [Result] Northouse L, Schafenacker A, Barr KL, Katapodi M, Yoon H, Brittain K, Song L, Ronis DL, An L. A tailored Web-based psychoeducational intervention for cancer patients and their family caregivers. Cancer Nurs. 2014 Sep-Oct;37(5):321-30. doi: 10.1097/NCC.0000000000000159. PMID 24945270